CLINICAL TRIAL: NCT04803630
Title: Survivor Warming to Alter Mood (S-WARM)
Brief Title: Thermal Therapy for the Treatment of Depression in Cancer Survivors, the S-WARM Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Awaiting grant funding for next phase of study
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 79318; NCI-2021-01102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 79318 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Hyperthermia, Induced; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment of depression (thermal therapy) (Experimental): Patients undergo thermal therapy over 2.5 hours.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Thermotherapy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Thermotherapy — Undergo thermal therapy
  Other Names: Heat Therapy

SUMMARY:
This early phase I trial evaluates the effect of thermal therapy on depression with or without sleep disturbance in cancer survivors. Thermal therapy may help improve quality of life, physical capacity, fatigue, and enhance positive mood and sleep quality. The purpose of this study is to evaluate the potential of thermal therapy to improve patient's quality of life by reducing symptoms of depression, sleep disruption, fatigue and anxiety in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the potential of thermal therapy to improve quality of life by reducing symptoms of depression in cancer survivors.

SECONDARY OBJECTIVE:

I. To evaluate the potential of thermal therapy to improve quality of life by reducing symptoms of sleep disruption in cancer survivors.

EXPLORATORY OBJECTIVE:

I. To evaluate the potential of thermal therapy to improve quality of life by reducing symptoms of fatigue, anxiety and other generally debilitating aspects of increased stress in cancer survivors.

OUTLINE:

Patients undergo thermal therapy over 2.5 hours.

After completion of study treatment, patients are followed up at weeks 1 or 2, 3 or 4, and then monthly for months 2-4.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had therapy for malignancy
* Age >= 18 years
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Patient denies current pregnancy
* Patients who screen positive on the depression/anxiety domain will be given the Hamilton Depression Rating Scale. Those with a score of 16 or more on this scale will be eligible for intervention

Exclusion Criteria:

* History of prior myocardial infarction. These patients may be allowed with clearance from a cardiologist
* History of any condition deemed by the principal investigator to be a contraindication to S-WARM therapy (e.g., skin reaction, dysregulation of thermoregulation, etc.)
* All patients with transdermal patches (e.g.; fentanyl, Lidoderm, scopolamine, etc.)
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive S-WARM
* Received an investigational agent within 30 days prior to enrollment
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2027-05-06 (Estimated)

PRIMARY OUTCOMES:
Change in depression | Baseline to 1 or 2 weeks after completion of therapy
  Measured by the Hamilton Depression Rating Scale.

SECONDARY OUTCOMES:
Durability of and variability in the response over time | Up to 4 months after completion of therapy
  Hypothesis tests of mixed effect model fixed effect slope parameters representing the population averaged changes in HDRS over time will be used to investigate whether the thermal intervention effects are durable over the course of the study.
Change in Pittsburgh Sleep Quality Index scores | Baseline, up to 4 months
  A 19 self-rated questionnaire. Each item is weighted on a 0-3 interval scale where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States